CLINICAL TRIAL: NCT00663312
Title: Impact of Deep Brain Stimulation of Subthalamic Nucleus on the Hepatic Glucose Production in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Pr Llorca, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0031
Record Dates: First submitted 2008-04-14; First posted 2008-04-22 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Idiopathic Parkinson's disease; Deep Brain stimulation; Hepatic glucose production; Insulin; Weight gain; Patient with an Idiopathic Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Insulin Resistance; Weight Gain | interventions — Proteins; Caloric Restriction

INTERVENTIONS:
Behavioral: e.g., Protein and calorie controlled diet; Self-hypnotic relaxation — Pilot description

SUMMARY:
Parkinson' disease is a neurodegenerative disorder characterised by bradykinesia, rigidity, rest tremor and postural instability. Dopaminergic therapy such as L-Dopa and dopamine agonists usually leads to a dramatic improvement of symptoms, but disease progression nevertheless remains inevitable. Bilateral Deep brain stimulation in subthalamic nucleus (STN) leads to a spectacular clinical improvement in patients with motor complications and is now considered as the gold standard surgical treatment.

However, this surgery induces a post-operative body weight gain which may limit the benefits of this technique and induce critical metabolic disorders such as profound alterations in the central control of energy metabolism. Previous data seems to show that glucose metabolism is also altered.

The aim of this prospective study was to identify if the STN stimulation could modify glucose metabolism regulation especially the endogen glucose production (by liver) Hypothalamus is able to detect glucose concentration variations and to control/adjust glucose levels by modulating the hepatic glucose production. As hypothamus and STN are anatomically closed, we hypothesise that the STN stimulation could modulate the hypothalamus function and consequently modify glucose production.

DETAILED DESCRIPTION:
ilot study 8 patients

Inclusion visit :

* Clinical examination/ Interview on health and medical history
* Complete UPDRS
* Body composition measured by DEXA
* Biologic check up
* MMS

Protocol :

All subjects were studied in the postabsorptive state after a 10-h overnight fast.

On the day of the experiment, patients do not receive their treatment (MED OFF). One catheter was retrogradely inserted into a dorsal vain and was used for blood sample. A second catheter was inserted into the controlateral arm for the tracer infusion. A continuous infusion of D-6,6 2H2 glucose (0,05mg/kg/h) was performed during 6 hours (after a primed dose of 0,05 mg/kg of this tracer).

The first 3 hours, patients were studied without stimulation (STIM OFF); the last 3 hours the stimulator was actuated (STIM ON). Blood samples were regularly collected for the 2H2 glucose enrichment determination, and for the insulin, glucose and glucagon plasma concentration analyses.

ELIGIBILITY:
Inclusion criteria :

* Age : 18-70 years
* Patient with an idiopathic Parkinson's disease according to the criteria of the "Parkinson's Disease Society Brain Bank" (Hughes et al., 1992)
* Patient treated with a deep brain stimulation according to the French consensus conference of treatment of Parkinson's disease (Consensus Conference Proceeding, 2000)
* Effect of the stimulation 50%
* Weight gain >5% (after surgery compared to before surgery)
* MMS>24/30
* No treatment modification 7 days before the inclusion
* Affiliation to social security
* Agreement of patients

Exclusion criteria :

* Patient treated with antibiotics, AINS, AIS or other treatment which could interfere with the protocol
* Patients with significant heart, respiratory, psychiatric, metabolic, hepatic, kidney diseases; diabetes, heart deficiency, chronic kidney deficiency, untreated thyroid disease …
* Patients with metabolic and/or biological anomalies
* Pregnant women
* Medical or chirurgical previous history which could interfere with the protocol
* Alcohol (>30g/day); Tobacco (>10 cigarettes/day)
* Participation to an other study at the same time

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the hepatic glucose production determined using the 2H2 glucose enrichment measurement and the infusion flow. | The hepatic glucose production was calculated during OFF stimulation period and ON stimulation period

SECONDARY OUTCOMES:
-Insulin plasma concentration kinetic -Glucose plasma concentration kinetic -Glucagon plasma concentration kinetic | During plasma concentration kinetic

CONTACTS AND LOCATIONS:
Overall Officials: Franck Durif, Pr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France

REFERENCES:
- [Derived] Batisse-Lignier M, Rieu I, Guillet C, Pujos E, Morio B, Lemaire JJ, Durif F, Boirie Y. Deep brain stimulation of the subthalamic nucleus regulates postabsorptive glucose metabolism in patients with Parkinson's disease. J Clin Endocrinol Metab. 2013 Jun;98(6):E1050-4. doi: 10.1210/jc.2012-3838. Epub 2013 Apr 30. PMID 23633215